CLINICAL TRIAL: NCT01037101
Title: D-Cycloserine as Enhancer of One-Session Treatment for Phobia of Heights in Adults
Brief Title: D-Cycloserine-Enhancer of One-Session Treatment for Phobia of Heights
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Collaborators: West Virginia University (Other); University of Charleston (Other)
Responsible Party: Principal Investigator, Crisitian Sirbu, PhD, Research Scientist, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-01-1896
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Height Phobia
Keywords: acrophobia; virtual reality; exposure therapy; In Vivo Exposure Therapy plus D-Cycloserine; In Vivo Exposure Therapy plus Placebo; Virtual Reality Exposure Therapy plus D-Cycloserine; Virtual Reality Exposure Therapy plus Placebo; Wait-List
MeSH Terms: conditions — Acrophobia | interventions — Virtual Reality Exposure Therapy; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- IVET+DCS (Active Comparator)
  Interventions: Behavioral: In Vivo Exposure Therapy; Drug: D-Cycloserine
- VRET+DCS (Experimental)
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Drug: D-Cycloserine
- VRET+Placebo (Experimental)
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Drug: Placebo
- IVET+Placebo (Active Comparator)
  Interventions: Behavioral: In Vivo Exposure Therapy; Drug: Placebo
- Wait-List (No Intervention): 3 weeks Wait-List

INTERVENTIONS:
Behavioral: In Vivo Exposure Therapy — Three hours of exposure therapy in a high place
  Arms: IVET+DCS; IVET+Placebo
Behavioral: Virtual Reality Exposure Therapy — Three hours of exposure therapy using a virtual reality system
  Arms: VRET+DCS; VRET+Placebo
Drug: D-Cycloserine — 50 mg of DCS administered 30 minutes before the session
  Other Names: Seromycin
  Arms: IVET+DCS; VRET+DCS
Drug: Placebo — 50 mg placebo administered 30 minutes before the session
  Arms: IVET+Placebo; VRET+Placebo

SUMMARY:
The study will determine the effects of D-Cycloserine (DCS) on fear reduction in patients diagnosed with phobia of heights (acrophobia) undergoing one session of three hours of virtual reality exposure therapy (VRET) or in vivo exposure therapy (IVET).

DETAILED DESCRIPTION:
The impact of D-Cycloserine on Virtual Reality Exposure Therapy (VRET) and In Vivo Exposure Therapy (IVET) for phobia of heights (acrophobia) will be tested using a randomized, double-blind, placebo-controlled trial. Eighty participants will be randomly assigned to one of the four treatment conditions: one-session VRET (3 hours) and 50 mg D-Cycloserine (VR-OST + DCS, N1=20); one-session VRET (3 hours) and placebo (VR-OST + Pl, N2=20); one-session IVET (3 hours) and placebo (IV + Pl, N3=20); or one-session IVET (3 hours) and 50 mg D-Cycloserine, (IV + DCS, N4=20). For twenty participants (5 from each group) the treatment will be delayed for three weeks and an additional assessment will be conducted as they will comprise a Wait List (WL) control group. Behavioral, cognitive and physiological changes in acrophobia will be assessed at pre-treatment, post-waitlist, post-treatment and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Men and women
* Diagnosis of acrophobia based on a clinical interview (ADIS-IV)
* Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

Exclusion Criteria:

* A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders; organic brain syndrome, cognitive dysfunction that could interfere with capacity to engage in therapy;
* A history of substance or alcohol dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the period of study participation.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate services.
* Patients must be off concurrent anxiolytics and beta blockers and on a stable dose of antidepressant medication for at least 3 weeks prior to initiation of randomized treatment.
* Patients receiving medication that might interfere with study medication (medication that might lower seizure threshold: meperidine or antibiotics in high dosage: penicillins, cephalosporins, amphotericin and imipenem),
* Patients with a current or past history of seizures
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted effective methods of contraception or abstinence
* Patients with a history of renal insufficiency (creatinine clearance less than 60 mL/min) or liver insufficiency
* Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration specifically targeting phobias
* Patients unable to understand study procedures and participate in the informed consent process.
* Other serious medical illnesses (e.g., cardiovascular, liver, kidney, respiratory, endocrine, neurologic, or blood-related diseases),
* Inability to tolerate wearing the Virtual Reality Head Mounted Display,
* If patients refuse the study medication
* Any allergic reactions to D-Cycloserine by history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Specific Phobia (acrophobia) diagnosis based on Anxiety Disorders Interview Schedule-IV (ADIS-IV) | One week post-treatment and 3 months folow-up

SECONDARY OUTCOMES:
Physiological responses to phobia-related stimuli, percentage of steps completed and Subjective Units of Distress during a Behavioral Avoidance Test (BAT) | One week post-treatment and 3 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Sirbu, Ph.D., Principal Investigator — CAMC Health System
Locations (1):
- West Virginia University School of Medicine Charleston Division, Charleston, West Virginia, United States